CLINICAL TRIAL: NCT03800277
Title: Prebiotic Supplementation and Metabolic Endotoxemia and Modulation of the Gut Microbiota: Double-blind and Randomized Parallel Clinical Study of the Efficacy and Synergistical Effect of Cranberry Polyphenols and Inulin From Agaves
Brief Title: Effect of Cranberry and Agaves Extract on Microbiota and Intestinal Health
Acronym: Phenulin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Ministry of Agriculture, Fisheries and Food, Quebec (Other Government); Ministry of economic development, innovation and export trade, Quebec (Unknown); Diana Food, Symrise (Unknown); Atrium Innovations (Industry); NutriAgaves, Mexico (Unknown); Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Principal Investigator, Helene Jacques, Professor, Laval University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GASTRO-Phenulin (2016-317)
Record Dates: First submitted 2018-12-06; First posted 2019-01-11 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Endotoxemia; Metabolic Syndrome; Glucose Metabolism Disorders; Insulin Resistance
MeSH Terms: conditions — Endotoxemia; Metabolic Syndrome; Glucose Metabolism Disorders; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cranberry and Agaves (Experimental): Cranberry extract (2 capsules) + Agaves powder (1 single-dose packet)
  Interventions: Dietary Supplement: Cranberry; Dietary Supplement: Agaves
- Cranberry and placebo (Experimental): Cranberry extract (2 capsules) + Placebo powder (1 single-dose packet)
  Interventions: Dietary Supplement: Cranberry; Dietary Supplement: Placebo
- Placebo and Agaves (Experimental): Placebo (2 capsules) + Agaves powder (1 single-dose packet)
  Interventions: Dietary Supplement: Agaves; Dietary Supplement: Placebo
- Placebo and placebo (Placebo Comparator): Placebo (2 capsules) + Placebo powder (1 single-dose packet)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Cranberry — Supplementation of polyphenols from cranberry extract
  Arms: Cranberry and Agaves; Cranberry and placebo
Dietary Supplement: Agaves — Supplementation of inulin from Agaves powder
  Arms: Cranberry and Agaves; Placebo and Agaves
Dietary Supplement: Placebo — Supplementation with placebo
  Arms: Cranberry and placebo; Placebo and Agaves; Placebo and placebo

SUMMARY:
The growing prevalence of obesity and type 2 diabetes (T2D) is a major public health problem. Recent studies have clearly established that the gut microbiota plays a key role in the investigator's propensity to develop obesity and associated metabolic health disorders. The gut microbiota compositions plays a decisive role in glucose metabolism and the chronic inflammatory state associated with insulin resistance. Consuming prebiotic rich diet, including polyphenol and inulin rich food could help modulate favorably the gut microbiota which could lead to a reduction of endotoxemia and beneficial metabolic health effects.

DETAILED DESCRIPTION:
It is now recognized that overweight individuals have altered microbiota which could lead to intestinal barrier defects and chronic inflammation disorders. Polyphenols such as Proanthocyanidins may modulate the gut microbiota thereby providing beneficial effects on metabolic health. Inulin is a well known prebiotic that could stimulate growth of favorable bacteria in the gut.

The overall goal is to determine the efficacy and synergy of a supplement of polyphenols from cranberry extract with or without a supplement of inulin from agaves to reduce chronic inflammation and endotoxemia and to improve glucose metabolism and insulin sensitivity by modulating microbiota of overweight human subjects with metabolic syndrome symptoms.

ELIGIBILITY:
Inclusion Criteria:

* overweight (BMI 25-39.9 kg/m2) or waist circumference ≥ 80 cm (women) and ≥94 cm (men)
* fasting insulin over 60 pmol/L or fasting glucose 5.6 - 6.9 mmol/L
* at least one of the following criteria: Tg ≥ 1.7 mmol/L; blood pressure ≥ 130/85 mmHg; HDL < 0,9 mmol/L; hsCRP 1-10 mg/L
* non-smoking
* eating fruits and vegetables less then 5 portions/day

Exclusion Criteria:

* chronic disease
* taking drugs or natural health products that could affect glucose or lipid metabolism
* taking anti-inflammatory, antiacids
* taking pre or probiotics
* inflammatory bowel disease
* antibiotics in the past 3 months
* allergy or intolerance to cranberries or agaves
* Major surgery in the past 3 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change in metabolic endotoxemia: Measure concentration of Lipopolysaccharides (LPS) and Lipopolysaccharide Binding Protein (LBP) in plasma | At the beginning and the end of treatment (10 weeks)
  effect of the supplements on variation in plasma concentration of LPS and LBP

SECONDARY OUTCOMES:
Change in intestinal permeability: Measure concentration of zonulin in plasma | At the beginning and the end of treatment (10 weeks)
  effect of the supplements on plasma concentration of zonulin
Change in inflammation state of the tissue: Measure concentration of calprotectin and lactoferrin in feces | At the beginning and the end of treatment (10 weeks)
  effect of the supplements on fecal calprotectin and lactoferrin
Change in systemic inflammation: Measure concentration of inflammation biomarkers in the serum | At the beginning and the end of treatment (10 weeks)
  effect of the supplements on chronic inflammation (serum concentration of hsCRP, Il-6, TNF-alpha, IL-1 beta, IL-23)
Change in glucose serum concentration | At the beginning and the end of treatment (10 weeks)
  effect of the supplements on serum concentration of glucose
Change in insulin and C-peptide serum concentration | At the beginning and the end of treatment (10 weeks)
  effect of the supplements on serum concentration of insulin and C-peptide
Change in microbiota diversity: growth of Akkermancia muciniphila, Lactobacillus, Prevotella, Bifdobacterium and inhibition of Clostridium perfringens, C. difficile, Bacteroides spp.) | At the beginning and the end of treatment (10 weeks)
  Global variation of the fecal microbiota and gut microbiota profiling

CONTACTS AND LOCATIONS:
Overall Officials: Hélène Jacques, PhD, Principal Investigator — Institute of nutrition and functional foods, Laval University; Yves Desjardins, PhD, Study Director — Institute of nutrition and functional foods, Laval University
Locations (1):
- Institute of nutrition and functional foods, Laval University, Québec, Quebec, Canada